CLINICAL TRIAL: NCT00620568
Title: An Ascending Multiple-Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of SLV-313 Sustained-Release (SR) Tablets Administered Orally to Subjects With Schizophrenia and Schizoaffective Disorder
Brief Title: Study Evaluating Multiple Ascending Dose in Schizophrenia Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3170A1-1001
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: SLV-313 SR
- 2 (Experimental)
  Interventions: Drug: SLV-313 SR
- 3 (Experimental)
  Interventions: Drug: SLV-313 SR
- 4 (Experimental)
  Interventions: Drug: SLV-313 SR

INTERVENTIONS:
Drug: SLV-313 SR — sustained release tablets taken once daily for 14 days

SUMMARY:
This is a randomized, inpatient, ascending multiple dose study to assess safety and tolerability of SLV-313 SR tablets administered orally to subjects with schizophrenia and schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged 18-50 years old
* Women, aged 18-50 years old

Exclusion Criteria:

* Non-lactating women, aged 18-50 years old
* Non-pregnant women, aged 18-50 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Observe safety and tolerability | 25 days

SECONDARY OUTCOMES:
PK and PD profile | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer